CLINICAL TRIAL: NCT05366634
Title: A Phase 1, Randomized, Placebo-controlled, Single-Blind, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MDK-703 in Healthy Adult Volunteers
Brief Title: A Single Ascending Dose Study to Evaluate MDK-703 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medikine, Inc. (Industry)
Collaborators: Medikine Australia Pty Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: MDK-703-101
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Single injection of MDK-703 (dose level 1) or matching placebo
  Interventions: Biological: MDK-703 or Placebo
- Cohort 2 (Experimental): Single injection of MDK-703 (dose level 2) or matching placebo
  Interventions: Biological: MDK-703 or Placebo
- Cohort 3 (Experimental): Single injection of MDK-703 (dose level 3) or matching placebo
  Interventions: Biological: MDK-703 or Placebo

INTERVENTIONS:
Biological: MDK-703 or Placebo — Injection

SUMMARY:
MDK-703-101 is a single ascending dose study, to determine the safety, tolerability, and PK/PD of MDK-703 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, autoimmune, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events after single injection of MDK-703 | 8 weeks
  Adverse events after single Injection

CONTACTS AND LOCATIONS:
Locations (1):
- Medikine Clinical Site, Herston, Queensland, Australia